CLINICAL TRIAL: NCT00385606
Title: Phase II-III, Factorial Multicenter Randomized Trial Evaluating the Addition of Rofecoxib to Polycht With Cispatin and Gemcitabine and Fixed Dose Rate Infusion of Gem in Association With Cisplatin in 1st-line for Advanced NSCLC
Brief Title: Study of Rofecoxib and Prolonged Constant Infusion of Gemcitabine in the Polychemotherapy Treatment of Advanced NSCLC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GECO
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2015-04

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: prolonged continuous infusion; Cox-2 inhibitors
MeSH Terms: interventions — Gemcitabine; Cisplatin; rofecoxib

ARMS (4):
- cisplatino plus gemcitabine (Active Comparator): Gemcitabina 1200 mg/m2 infusion of 30 minutes at day 1, 8 + cisplatin 80 mg/m² day 1, every 3 weeks for 6 cycles.
  Interventions: Drug: gemcitabine; Drug: cisplatin
- cisplatino plus gemcitabine plus rofecoxib (Experimental): Gemcitabina 1200 mg/m2 infusion of 30 minutes at day 1, 8 + cisplatin 80 mg/m² day 1, every 3 weeks + rofecoxib 50 mg/die per os until progression of disease.
  Interventions: Drug: gemcitabine; Drug: cisplatin; Drug: rofecoxib
- cisplatino plus gemcitabine 10 mg/m2/min (Experimental): Gemcitabina 1200 mg/m2 infusion of 120 minutes at day 1, 8 + cisplatin 80 mg/m² day 1, every 3 weeks for 6 cycles.
  Interventions: Drug: prolonged continuous infusion gemcitabine; Drug: cisplatin
- cisplatino plus gemcitabine 10 mg/m2/min plus rofecoxib (Experimental): Gemcitabina 1200 mg/m2 infusion of 120 minutes at day 1, 8 + cisplatin 80 mg/m² day 1, every 3 weeks + rofecoxib 50 mg/die per os until progression of disease.
  Interventions: Drug: prolonged continuous infusion gemcitabine; Drug: cisplatin; Drug: rofecoxib

INTERVENTIONS:
Drug: gemcitabine
  Arms: cisplatino plus gemcitabine; cisplatino plus gemcitabine plus rofecoxib
Drug: prolonged continuous infusion gemcitabine
  Arms: cisplatino plus gemcitabine 10 mg/m2/min; cisplatino plus gemcitabine 10 mg/m2/min plus rofecoxib
Drug: cisplatin
Drug: rofecoxib
  Arms: cisplatino plus gemcitabine 10 mg/m2/min plus rofecoxib; cisplatino plus gemcitabine plus rofecoxib

SUMMARY:
The purpose of this study is to evaluate the tolerability and efficacy of the addition of rofecoxib to first-line chemotherapy, and to evaluate the efficacy of prolonged continuous infusion of gemcitabine in combination with cisplatin in the treatment of patients affected by advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
The primary end-points of the GECO study

* To evaluate the tolerability of three innovative schedules of treatment for advanced NSCLC
* To evaluate the efficacy of the addition of rofecoxib to first-line chemotherapy in the treatment of patients affected by advanced NSCLC
* To evaluate the efficacy of prolonged continuous infusion (p.c.i.) of gemcitabine, with the fixed infusion rate of 10 mg/sqm/minute) versus the standard administration in 30 minutes, in combination with cisplatin, in the treatment of patients affected by advanced NSCLC

Four treatment arms are planned.

* ARM A standard treatment : cisplatin + gemcitabine
* ARM B cisplatin + gemcitabine + rofecoxib
* ARM C cisplatin + p.c.i. gemcitabine (10 mg/sqm/minute)
* ARM D cisplatin + p.c.i gemcitabine (10 mg/sqm/minute) + rofecoxib

The phase II part of the study for experimental arms B, C and D will be conducted to evaluate tolerability in the three treatment arms.

The phase III study for efficacy has been designed according to a factorial 2x2 model with the planned comparison of

* The efficacy of rofecoxib: A + C (arms without rofecoxib) vs B+D (arms with rofecoxib)
* The efficacy of p.c.i. gemcitabine: A + B (arms with standard infusion of gemcitabine) vs C+ D (arms with p.c.i gemcitabine)

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic diagnosis of non-small cell lung cancer
* Disease stage IIIB or IV
* Age less than 70 years
* ECOG performance status 2 or less
* Patients with cerebral metastases are permitted if they are asymptomatic and do not require radiation therapy concomitant with chemotherapy
* Negative history of allergy to non-steroidal anti-inflammatory and/or sulphonamide drugs
* Patients previously treated with radiation therapy are permitted if at least 4 weeks have passed since last therapy
* Written informed consent

Exclusion Criteria:

* Previous chemotherapy
* Previous or concomitant malignant neoplasm (excluding adequately treated baso or spinocellular skin carcinoma or carcinoma in situ of the cervix)
* Neutrophil < 2000/mm3, platelets < 100,000/mm3, haemoglobin < 10 g/dl
* Creatinine > 1.25 x the upper normal limits
* GOT and/or GPT and/or Bilirubin > 1.25 the upper normal limits in absence of hepatic metastases
* GOT and/or GPT and/or Bilirubin > 2.5 the upper normal limits in presence of hepatic metastases
* Any concomitant pathology that would, in the investigator's opinion, contraindicate the use of the drugs in this study
* Inability to comply with follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2003-01; Primary Completion 2005-12 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the tolerability of three experimental treatment schedules | at the end of each cycle of chemotherapy (every 3 weeks) until 21 days after the last treatment administrationministration
  adverse events according to CTCAE criteria
To evaluate the efficacy of the addition of rofecoxib to first-line chemotherapy | at the end of cycle 3 and cycle 6 until the date of first documented PD (up to 1 year).
  response rate according to RECIST criteria
To evaluate the efficacy of prolonged continuous infusion (p.c.i.) of gemcitabine vs standard infusion, in combination with cisplatin | at the end of cycle 3 and cycle 6 until the date of first documented PD (up to 1 year).
  response rate according to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — San Giuseppe Moscati Hospital, Avellino, Italy; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute Naples, Italy
Locations (25):
- Italy (25):
  - Azienda Ospedaliera S. Giuseppe Moscati, U.O. di Oncologia Medica, Monteforte Irpino, AV
  - Ospedale Regionale Miulli, Divisione Medicina Interna Sezione Oncologica, Acquaviva delle Fonti, BA
  - IRCCS Oncologico Bari, Oncologia Medica, Bari, BA
  - Istituto Oncologico di Bari, U.O. di Oncologia Medica e Sperimentale, Bari, BA
  - Policlinico Universitario, Oncologia Medica II, Cagliari, CA
  - Ospedale A. Cardarelli, Campobasso, CB
  - Ospedale Mariano Santo, U.O. di Oncologia Medica, Cosenza, CS
  - Ospedale Umberto di Frosinone, Frosinone, FR
  - Ospedale Civile di Legnano, Legnano, MI
  - Ospedale S. Paolo, Milan, MI
  - Policlinico Universitario P. Giaccone, Palermo, PA
  - Casa di Cura La Maddalena S.p.A., Dipartimento Oncologico, Palermo, PA
  - Istituto Oncologico Veneto, Padua, PD
  - Ospedale Civile Umberto I, Day Hospital Oncoematologico, Nocera Inferiore, SA
  - Divisione di Oncologia Medica, U.S.L.L. 13, Noale, VE
  - Ospedale S. Bortolo ULSS 6, U.O. di Oncologia Medica, Vicenza, VI
  - Ospedale L. Sacco, Milan
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli
  - Istituto Nazionale dei Tumori, Divisione di Oncologia Medica C, Napoli
  - Second University of Naples, Napoli
  - Ospedale Santa Corona, Pietre Ligure
  - Istituto Regina Elena, Divisione di Oncologia Medica, Roma
  - Ospedale S. Giovanni Calibita Gatebenefratelli, Roma
  - Ospedale San Camillo - Forlanini, Rome
  - Azienda Ospedaliera Di Busto Arsizio, Saronno

REFERENCES:
- [Result] Gridelli C, Gallo C, Ceribelli A, Gebbia V, Gamucci T, Ciardiello F, Carozza F, Favaretto A, Daniele B, Galetta D, Barbera S, Rosetti F, Rossi A, Maione P, Cognetti F, Testa A, Di Maio M, Morabito A, Perrone F; GECO investigators. Factorial phase III randomised trial of rofecoxib and prolonged constant infusion of gemcitabine in advanced non-small-cell lung cancer: the GEmcitabine-COxib in NSCLC (GECO) study. Lancet Oncol. 2007 Jun;8(6):500-12. doi: 10.1016/S1470-2045(07)70146-8. PMID 17513173
- [Derived] Di Maio M, Gallo C, Leighl NB, Piccirillo MC, Daniele G, Nuzzo F, Gridelli C, Gebbia V, Ciardiello F, De Placido S, Ceribelli A, Favaretto AG, de Matteis A, Feld R, Butts C, Bryce J, Signoriello S, Morabito A, Rocco G, Perrone F. Symptomatic toxicities experienced during anticancer treatment: agreement between patient and physician reporting in three randomized trials. J Clin Oncol. 2015 Mar 10;33(8):910-5. doi: 10.1200/JCO.2014.57.9334. Epub 2015 Jan 26. PMID 25624439